CLINICAL TRIAL: NCT03885063
Title: Modifying a Telephone Based Care Program to Assess for Self-Neglect
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic interrupted study proceudres
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Constance Johnson, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSC-SN-18-0741
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Self Neglect

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benjamin Rose Institute Care Consultation (BRI-CC) (Experimental)
  Interventions: Behavioral: Benjamin Rose Institute Care Consultation (BRI-CC)
- No intervention (No Intervention)

INTERVENTIONS:
Behavioral: Benjamin Rose Institute Care Consultation (BRI-CC) — The BRI-CC is a telephone-based intervention designed for adults with chronic conditions and has been used in persons with dementia and their caregiver (CG). This assessment is guided by the use of assessment tools with domains that trigger specific and pertinent needs of the dyad such as relationship strain, depression, financial concerns, memory problems, and difficult behaviors. To address unmet needs, the care consultant and dyad develop action plans with specific action steps pertinent to the dyad. The intervention involves maintenance and support where the care consultant (CC) continues the relationship with the dyad through regular telephone contact, email and mail. CC use a web-based reporting system, to maintain and track dyad information, assessments, action plans, completed tasks, and ongoing contacts. At a minimum, the care consultant will contact the dyad by telephone once per month over the duration of the study period (i.e. 6 months).
  Arms: Benjamin Rose Institute Care Consultation (BRI-CC)

SUMMARY:
The purpose of this study is to assess the feasibility of enrollment, attrition, and adherence of Benjamin Rose Institute Care Consultation (BRI-CC) on unmet needs in low-income older adults who screen positive for dementia and their caregiver (CG).

ELIGIBILITY:
Inclusion Criteria:

* able to provide consent and understand English since most of the measures have not been translated into other languages
* has a CG willing to participate, specifically the CG must provide assistance in personal care, daily living tasks, and/or healthrelated decisions at least 3 hours per day and at least 3 days per week
* screen positive for dementia.

Exclusion Criteria:

* participant who receives home-delivered meals plans to relocate to long-term care prior to study enrollment
* reportedly moving out of the catchment area during the proposed study period
* non-English speaking
* unable to provide informed consent
* pre-diagnosed terminal illness
* non-working telephone
* visual impairment inhibiting the dyad from reading the instruments

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Feasibility as assessed by enrollment rate | 6 months
  enrollment rate = # enrolled / # who met inclusion criteria
Feasibility as assessed by attrition rate | 6 months
  attrition rate = # not completing the study
  / # enrolled at baseline
Feasibility as assessed by adherence rate | 6 months
  adherence rate = # completing all BRI-CC sessions / # enrolled in intervention group
Feasibility as assessed by why subjects were not able to participate in BRI-CC | 6 months
Feasibility as assessed by why subjects dropped out of BRI-CC | 6 months

SECONDARY OUTCOMES:
Unmet needs of participants who receive home-delivered meals as assessed by domains of the Unmet Needs Instrument | baseline
  Responses will be entered onto a 10-item dichotomous response (need met or unmet) instrument that will be summed across six assessment domains: 1) understanding dementia, 2) accessing healthcare services, 3) accessing community services 4) accessing family services, 5) legal and financial issues, and 6) emotional support.
Unmet needs of of participants who receive home-delivered meals as assessed by domains of the Unmet Needs Instrument | 3 months
  Responses will be entered onto a 10-item dichotomous response (need met or unmet) instrument that will be summed across six assessment domains: 1) understanding dementia, 2) accessing healthcare services, 3) accessing community services 4) accessing family services, 5) legal and financial issues, and 6) emotional support.
Unmet needs of participants who receive home-delivered meals as assessed by domains of the Unmet Needs Instrument | 6 months
  Responses will be entered onto a 10-item dichotomous response (need met or unmet) instrument that will be summed across six assessment domains: 1) understanding dementia, 2) accessing healthcare services, 3) accessing community services 4) accessing family services, 5) legal and financial issues, and 6) emotional support.
Self Neglect as assessed by the Elder Self-Neglect Instrument (of participants who receive home-delivered meals) | baseline
  The Elder Self-Neglect Assessment (ESNA) is a 25-item rating scale to assess for SN.
  Each item is a 5-point Likert scale to assess the participant and the participant's home. Scores are tallied with the following suggested interpretations: (1) if high scores for social behavioral SN (B) but not environmental SN (E), then there is high risk for SN, (2) if high scores are for both B & E, then severe unintentional SN, and (3) if high E but not B, then intentional SN. An item example asks, "Does the older adult wear dirty clothes"?
Self Neglect as assessed by the Elder Self-Neglect Instrument (of participants who receive home-delivered meals) | 6 months
  The Elder Self-Neglect Assessment (ESNA) is a 25-item rating scale to assess for SN. Each item is a 5-point Likert scale to assess the participant and the participant's home. Scores are tallied with the following suggested interpretations: (1) if high scores for social behavioral SN (B) but not environmental SN (E), then there is high risk for SN, (2) if high scores are for both B & E, then severe unintentional SN, and (3) if high E but not B, then intentional SN. An item example asks, "Does the older adult wear dirty clothes"?
Number of participants who receive home-delivered meals who were admitted to the hospital | 6 months
Number of participants who receive home-delivered meals who were readmitted to the hospital | 6 months
Number participants who receive home-delivered meals who were relocated for long term care | 6 months
Psychosocial well-being of the caregiver (CG) as assessed by the Zarit Burden Interview | baseline
  The Zarit Burden Interview is a 22-item self-rated screen to assess CG burden. This measure uses a 5-point Likert scale to assess direct stress of the CG, specifically caregivers of persons with dementia. It has been shown to be sensitive to change.
Psychosocial well-being of the informal caregiver as assessed by the Zarit Burden Interview | 6 months
  The Zarit Burden Interview is a 22-item self-rated screen to assess CG burden. This measure uses a 5-point Likert scale to assess direct stress of the CG, specifically caregivers of persons with dementia. It has been shown to be sensitive to change.
Caregiver depression as assessed by the Geriatric Depression Scale- Short Form | baseline
  The Geriatric Depression Scale (Short-Form) (GDS-SF) is a 15-item "yes" and "no" self-rated screen to assess depression. Scores range from 0-15 with scores of 5 and greater are indicative of depression
Caregiver depression as assessed by the Geriatric Depression Scale- Short Form | 6 months
  The Geriatric Depression Scale (Short-Form) (GDS-SF) is a 15-item "yes" and "no" self-rated screen to assess depression. Scores range from 0-15 with scores of 5 and greater are indicative of depression
Caregiver unmet needs as assessed by domains of the Unmet Needs Instrument | baseline
  Responses will be entered onto a 10-item dichotomous response (need met or unmet) instrument that will be summed across six assessment domains: 1) understanding dementia, 2) accessing healthcare services, 3) accessing community services 4) accessing family services, 5) legal and financial issues, and 6) emotional support.
Caregiver unmet needs as assessed by domains of the Unmet Needs Instrument | 6 months
  Responses will be entered onto a 10-item dichotomous response (need met or unmet) instrument that will be summed across six assessment domains: 1) understanding dementia, 2) accessing healthcare services, 3) accessing community services 4) accessing family services, 5) legal and financial issues, and 6) emotional support.
Emotional significance of pets to participants who receive home-delivered meals as assessed by the Monash Dog Owner Relationship Scale (MDORS) | baseline
Unmet Pet Care needs of participants who receive home-delivered meals as assessed by the Unmet Pet Care Needs (UPCN) scale | baseline
  The UPCN scale was developed by the researchers which taps a respondent's need for information or help surrounding pet-related issues. It is based on the Benjamin Rose Institute Unmet Needs Scale (see references). Response categories are dichotomous (0=No and
  1=Yes). The total score is the sum of the items noted for each measure. Higher scores indicate greater unmet need for information or help. The individual scales may be summed to create a score for total unmet need.
Barriers to pet caretaking as assessed by structured interviews over the telephone with participants who receive home-delivered meals | baseline
Potential resources and services to support unmet pet caretaking needs as assessed by structured interviews over the telephone with participants who receive home-delivered meals | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Pickens, PhD, RN, MSN, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No